CLINICAL TRIAL: NCT02971098
Title: Novel Molecular Mechanisms of Skeletal Muscle Insulin, Resistance if Physically Inactive Older Adults
Brief Title: Mechanisms of Skeletal Muscle Insulin Resistance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Ph.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 84354
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Reduced Physical Activity

STUDY DESIGN:
Intervention Model Description: 2 weeks of physical inactivity
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced activity (Experimental): participants will undergo a reduced physical activity period (75% step reduction) for two weeks.
  Interventions: Procedure: Reduced activity

INTERVENTIONS:
Procedure: Reduced activity — Participants will reduced their physical activity level to approximately 2000 steps or 75% of their normal activity levels.

SUMMARY:
The over-65 population is not only increasing at an alarming rate, but because six out of 10 will be managing more than one chronic condition by 2030, they will make up a much greater proportion of hospitalizations than ever before. Hospitalizations for disease, injury, and/or surgery in this group are likely to impair physical mobility and, therefore, the older adults capacity to be physically active both during hospitalization and beyond. The resulting sedentary lifestyle is likely to be accepted as the "new normal", ultimately increasing the risk of skeletal muscle and metabolic dysfunction (e.g. impaired glucose disposal, insulin resistance). These devastating outcomes are neither inevitable nor necessary if prevented with an appropriate mechanism-based intervention.

A novel mechanism that may contribute to physical inactivity-induced insulin resistance is accumulation of inflammation and ceramide within skeletal muscle. Of interest, increased skeletal muscle inflammation and ceramide has been tied to various metabolic disturbances such as diabetes and insulin resistance. However, it is currently unknown if skeletal muscle inflammation and ceramide are a key mechanism associated with insulin resistance due to physical inactivity in older adults.

DETAILED DESCRIPTION:
The investigator team will recruit younger and older (N=8; 18-35y and 60-85 yrs) male and female adults recruited in the Salt Lake City area.

The investigator team will then schedule separate visits for Strength, Power and Physical Function and the separate visits for Lean Mass and OGTT measurements (see description below).

1. Lean Mass, oral glucose tolerance test , Strength, Power, Exercise Testing and Physical Function Measurements. Lean mass assessment via dual-energy X-ray absorptiometry (DXA), ultra sound and peripheral quantitative computed tomography (pQCT) will be assessed in the center for clinical and translational sciences (CCTS) while knee extensor isometric strength, power and physical function testing will be conducted in the Skeletal muscle exercise research facility (SMERF) laboratory (520 Wakara Way). These endpoints will be considered secondary objectives to determine relationships with insulin sensitivity and muscle cell signaling events. These tests will occur within one week before the reduced activity experiment and will be repeated after completing the reduced activity period and after exercise training. For lean mass assessment, subjects will be tested in the morning after an overnight fast prior to the DXA scan. Isometric strength will be assessed in both legs with a maximal voluntary isometric contraction effort (at a 600 knee angle) developed by the knee extensors (quadriceps) and plantar/dorsi flexor muscles on a dynamometer. For lower extremity extension power testing a Nottingham power rig will be used. The following battery of functional performance tests will be used: Stair ascent/descent time, six-minute walk distance, 50 foot walk time, and the timed up and go test. All tests are tests that we frequently and safely perform in older individuals.

   Maximal oxygen consumption (exercise testing) will be measured by a metabolic cart during a graded maximal exercise test on a stationary cycle ergometer. This test will be performed in the CCTS under direct supervision of an exercise physiologist.
2. Physical Activity Monitoring, Dietary Record. Subjects will be fitted with an ankle Step Activity Monitor in order to determine their daily level of physical activity over 7 days period preceding the reduced physical activity study. Additionally, a 3-day daily dietary record will be self-reported before this period. The participant will be properly instructed by a research team member on how to conduct this reporting and how to wear the ankle activity monitor.
3. Insulin Clamp Study, Metabolic Rate and Muscle Biopsies. On a separate day, participants will arrive at the CCTS fasted in the morning on Day 1 and a euglycemic-hyperinsulinemic clamp study will be performed as we have done previously. The research team physician will oversee the clamp procedure as he is very experienced using this method.

   Metabolic rate will be determined 30 minutes before the initiation of the insulin infusion and 30 minutes at the end of the insulin infusion period. Metabolic rate will be determined using a indirect calorimeter housed at the CCTS. To do so, the participant will be fitted with a canopy hood. The participant with breathe normally for 30 minutes during the procedure. The canopy will be removed then the first muscle biopsy will occur.

   A vastus lateralis muscle biopsy will be sampled before and 3h after the clamp combined with periodic blood sampling for measure of fasting and insulin-stimulated insulin, glucose, muscle cell signaling endpoints, and specific ceramide species. Biopsies will occur on opposite legs. Muscle biopsies were be performed by trained CCTS nurses as we have done routinely in our bed rest studies in older adults. Muscle samples will then be flash-frozen in liquid nitrogen and stored for later analysis. After the clamp experiment, subjects will begin the reduced physical inactivity study which will take place at the participant home.

   On Day 14, the participant again will return to the CCTS following an overnight fast and the insulin clamp study will be repeated in order to make comparisons to the pre insulin clamp study (Day 1).
4. Reduced Physical inactivity experiment. After completion of the first insulin clamp experiment (Day 1), subjects will adhere to 14-days of reduced physical activity at their home as has been conduced before. The goal will be for the participant to maintain no more than ~2000 steps/day as determined by a monitor that the subject will be able to see and record. The investigators will inform the participant that their normal diet should remain the same. As mentioned above, on day 7, the participant will return for a DXA scan, OGTT's and thigh muscle biopsies. Also mentioned above, on Day 14, after an overnight fast, a second insulin clamp study coupled with muscle biopsies will be conducted as detailed above in the CCTS. Lean mass, strength, power, and physical function measurements will be re-assessed on a later day following the reduced activity study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-85 yrs
* Ability to sign informed consent
* Free-living, prior to admission

Exclusion Criteria:

* The participant must not have participated in any previous research studies utilizing ionizing radiation (either radioisotopes or diagnostic x-rays) during the past 12 months in order to participate in this study. Cardiac abnormalities considered exclusionary by the study physician
* Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
* History of kidney disease or failure
* Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
* Risk of deep vein thrombosis (DVT) including family history of thrombophilia, DVT, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocysteinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombin III
* Use of anticoagulant therapy (e.g., Coumadin, heparin)
* Elevated systolic pressure >150 or a diastolic blood pressure > 100
* Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Currently on a weight-loss diet or body mass index > 30 kg/m2
* Recent anabolic or corticosteroids use (within 3 months)
* History of stroke with motor disability
* A recent history (<12 months) of GI bleed
* Exercise training (>2 session of moderate to high intensity aerobic or resistance exercise/week)
* History of liver disease
* History of respiratory disease (acute upper respiratory infection, history of chronic lung disease)
* Prior history of Heparin-Induced Thrombocytopenia (HIT)
* Any other condition or event considered exclusionary by the PI and faculty physician
* An HbA1c value at or greater than 6.5%
* Subjects may not participate if they have utilized ionizing radiation (either radioisotopes or diagnostic x-rays) during the past 12 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Steady state glucose infusion rate | percent change from baseline at 14 days
  Glucose infusion rate will be determined by a hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
lean mass | percent change from baseline at 14 days
  lean mass will be determined by DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Micah J Drummond, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No